CLINICAL TRIAL: NCT05740553
Title: Using the ReTrieve Automated Stereognosis System to Treat Loss of Tactile Function After Brain Injury
Brief Title: Automated Stereognosis to Treat Loss of Tactile Function After Brain Injury
Acronym: ReTrieve
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate participant recruitment (potentially due to COVID-19)
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-12
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-01

CONDITIONS: Stroke; Chronic Brain Injury; Peripheral Neuropathy
MeSH Terms: conditions — Stroke; Brain Injury, Chronic; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participants complete tactile training for 6-8 weeks, and complete no additional training for 8 weeks. One group will begin with tactile training, and the other group will begin with no additional training, then they will swap. At each time point (before portion 1, after portion 1, and after portion 2) their tactile function will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training First (Experimental)
  Interventions: Device: ReTrieve Automated Stereognosis System
- Training Second (Experimental)
  Interventions: Device: ReTrieve Automated Stereognosis System

INTERVENTIONS:
Device: ReTrieve Automated Stereognosis System — An automated tactile training system that may help patients recover lost tactile function after brain injury.

SUMMARY:
Researchers aim to determine whether the ReTrieve system for tactile training can improve tactile function (sense of touch) in the hand after brain injury when used at home for 6 weeks.

DETAILED DESCRIPTION:
All participants who have been found eligible for this study and given informed consent will be randomized into two groups- either participants will begin ReTrieve training immediately following an initial assessment, or wait 8 weeks before beginning training.

During the study, participants will have a ReTrieve tactile training system delivered home for use over 6 weeks. Investigators will take three days to teach participants how to use the system. Each week for the remainder of the 6 weeks, participants will use this system for 4+ days per week on their own, and for 1 day supervised. During each supervised day, participants will complete approximately 1 hour of training while supervised over video chat with researchers.

Participants' tactile function will be assessed at three separate time points: once within one week before beginning training, once within one week after completing training, as well as once either 8 weeks before or 8 weeks after the training. This assessment has a required survey component, as well as an optional in-person clinical assessment component.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Be able to communicate and consent for themselves
* Have experienced a brain injury more than 6 months prior to the date of study participation
* Have chronic tactile deficits in at least one hand as a result of their brain injury
* Have sufficient motor ability in their affected hand(s) to complete reach and grasp tasks
* Have sufficient motor ability in their affected hand(s) to raise their arms above their head
* Have sufficient motor ability in their affected hand(s) to hold objects
* Have wireless internet and a laptop or mobile device at home for video conferencing
* Live in the greater Dallas area

Exclusion Criteria:

* Significant cognitive deficits that would preclude them from understanding instructions
* Significant communication deficits that would preclude them from consenting for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Number of Retrievals | 6-8 weeks
  The majority of participants should manage at least 4500 retrievals over their ~30 hours of system use
Number of Retrievals per Hour | 6-8 weeks
  The majority of participants should achieve at least 700 retrievals per hour by the end of training

SECONDARY OUTCOMES:
Improved Tactile Function | 6-8 weeks
  Participants should show a significantly greater increase in tactile function as measured by the French variation of the Upper Extremity subscore of the Erasmus modified Nottingham Sensory Assessment [High scores are better. Assessment performed for both hands. Scores range from 0-48 (0-24 per hand) on somesthesia, and 0-20 (0-10) on stereognosis. Total score range per participant is 0-68 (0-34 per hand)] when measured over their 6-8 weeks of tactile training than when measured over their 8 weeks without tactile training.
Improved Perceived Tactile Function | 6-8 weeks
  Participants should show a significantly greater increase in their perceived tactile function score as measured by the 'ABILHAND' questionnaire [High scores are better. Answered for only most impaired hand. 23 activities scored 0(impossible)-2(easy) Score range 0-46] combined with a modified version of the Sensory Perception Quotient (modified to focus on tactile and remove temperature) [High scores are better. Score range 0-18. Answered for only most impaired hand.] when measured over their 6-8 weeks of tactile training than when measured over their 8 weeks without tactile training.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided